CLINICAL TRIAL: NCT05953987
Title: Effects of Aerobic Combined With Diaphragmatic Breathing Exercise on Pulmonary Function, Smoking Cessation, and Urine Cotinine Among Smokers
Brief Title: Effects of Aerobic Combined With Diaphragmatic Breathing Exercise in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 7
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Smoker Lung; Smoking Cessation
Keywords: Smoker; Aerobic exercise; Respiratory muscle strength
MeSH Terms: conditions — Smoking Cessation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Twenty-four smokers aged between 20 and 45 years were allocated into 3 groups: a sedentary control group (CON, n = 8), an aerobic exercise group (EX, n = 8), and an aerobic combined with diaphragmatic breathing exercise group (EXDB, n = 8). The general physiological characteristics, pulmonary function, and respiratory muscle strength values before and after 8 weeks were meas-ured. The Quit Smoking Questionnaire and urine cotinine were measured for either 30 days after the training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic combined with diaphragmatic breathing exercise (EXDB) (Experimental): The participant underwent diaphragmatic breathing exercises which were performed in a supine position, gradually in-creasing the weight by 2.5 kg in weeks 1-4 and further increasing to 5 kg in weeks 5-8. After completing the prescribed breathing exercises and taking a 60-second rest, participants proceeded to perform aerobic exercises, either by running on a treadmill or on a regular floor surface. Each training session began with a 5-minute warm-up comprising stretching exercises. In weeks 1-4, moderate intensity was maintained, targeting 40-50% of the heart rate reserve (HRR) for a duration of 60 minutes. From weeks 5-8, the intensity increased to the range of 51-60% of the heart rate reserve, and a 5-minute cool down was added.
  Interventions: Other: aerobic combined with diaphragmatic breathing exercise (EXDB)
- aerobic exercise (EX) (Experimental): The participant underwent aerobic exercises, either by running on a treadmill or on a regular floor surface. Each training session began with a 5-minute warm-up comprising stretching exercises. In weeks 1-4, moderate intensity was maintained, targeting 40-50% of the heart rate reserve (HRR) for a duration of 60 minutes. From weeks 5-8, the intensity increased to the range of 51-60% of the heart rate reserve, and a 5-minute cool down was added.
  Interventions: Other: aerobic exercise (EX)
- sedentary control (CON) (Other): The participant did not engage in the aerobic exercise training protocol or receive any form of supplementation during the study trial.
  Interventions: Other: sedentary control (CON)

INTERVENTIONS:
Other: aerobic combined with diaphragmatic breathing exercise (EXDB) — The participant underwent diaphragmatic breathing exercises which were performed in a supine position, gradually in-creasing the weight by 2.5 kg in weeks 1-4 and further increasing to 5 kg in weeks 5-8. After completing the prescribed breathing exercises and taking a 60-second rest, participants proceeded to perform aerobic exercises, either by running on a treadmill or on a regular floor surface. Each training session began with a 5-minute warm-up comprising stretching exercises. In weeks 1-4, moderate intensity was maintained, targeting 40-50% of the heart rate reserve (HRR) for a duration of 60 minutes. From weeks 5-8, the intensity increased to the range of 51-60% of the heart rate reserve, and a 5-minute cool down was added
  Arms: aerobic combined with diaphragmatic breathing exercise (EXDB)
Other: aerobic exercise (EX) — The participant underwent aerobic exercises, either by running on a treadmill or on a regular floor surface. Each training session began with a 5-minute warm-up comprising stretching exercises. In weeks 1-4, moderate intensity was maintained, targeting 40-50% of the heart rate reserve (HRR) for a duration of 60 minutes. From weeks 5-8, the intensity increased to the range of 51-60% of the heart rate reserve, and a 5-minute cool down was added.
  Arms: aerobic exercise (EX)
Other: sedentary control (CON) — The participant did not engage in the aerobic exercise training protocol or receive any form of supplementation during the study trial.
  Arms: sedentary control (CON)

SUMMARY:
This study aimed to evaluate the effectiveness of aerobic exercise combined with diaphragmatic breathing exercise on pulmonary function and smoking cessation among smokers.

DETAILED DESCRIPTION:
Twenty-four smokers aged between 20 and 45 years were allocated into 3 groups: a sedentary control group (CON, n = 8), an aerobic exercise group (EX, n = 8), and an aerobic combined with diaphragmatic breathing exercise group (EXDB, n = 8). The general physiological characteristics, pulmonary function, and respiratory muscle strength values before and after 8 weeks were meas-ured. The Quit Smoking Questionnaire and urine cotinine were measured for either 30 days after the training.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals included those who set the quit date within 7 days from the date of calling the TNQ. The participants have smoked more than or equal to 10 cigarettes per day for at least 1 year and had a body mass index of not more than 24.9 kg/m2. More-over, they were screened for the health risks of exercise by the Physical Activity Readiness Questionnaire (PAR-Q). They must not have exercised for 30 minutes or more at least three times a week for the past six months.

Exclusion Criteria:

* This study excluded participants with a history of respiratory system diseases such as pulmonary tuberculosis, asthma, chronic obstructive pulmonary disease, lung cancer, etc. and who were using nicotine replacement therapy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | Change from Baseline pulmonary function at 8 weeks.
  The anticipated value and liters of FVC, FEV1, and MVV maneuver were measured using a computerized spirometer (SpirobankG) in accordance with the pulmonary function test criteria of the American Thoracic Society. Participants were asked to sit on a chair with a nasal clip on. Before demonstrating forced inspiration and expiration and returning to normal breathing, three cycles of slow normal breathing were performed. Participants were instructed to inhale and exhale quickly and strongly for 15 seconds during the MVV maneuver.
Smoking cessation | Change from Baseline Smoking cessation at 8 weeks, and 12 weeks
  The Quit Smoking Questionnaire was utilized to evaluate the smoking status of each participant by posing the following question: "Did you refrain from smoking continuously for a minimum of 7 days after your designated quit date?" If the response was affirmative, the participants were further inquired about their continuous abstinence for either 30 days after the training. Four items within the questionnaire yielded a Cronbach's alpha coefficient of 0.93
Urine cotinine | Change from Baseline Urine cotinine at 8 weeks, and 12 weeks
  The Direct Barbituric Acid (DBA) reaction method was utilized to measure urine cotinine. The results were interpreted based on the color change observed in the urine sample. Each morning, a urine sample of 30-50 ml was collected and added to the urinary cotinine measurement kit by participants. The color of the sample was then com-pared to the standard color band for urinary cotinine, and pictures were taken to be sent to the researchers. Assessment was conducted at 30 days after training, and the results were categorized as either "found" or "not found" based on the color change observed in the test tabs

SECONDARY OUTCOMES:
Respiratory muscle strength | Change from Baseline Respiratory muscle strength at 8 weeks.
  A portable handheld mouth pressure meter (Micro RPM England) was used to test respiratory muscle strength. For the MIP assessment, participants were told to exhale until they felt no air remaining in their lungs (starting at the functional residual capacity [FRC]). They then inhaled for 1-2 seconds while holding the item in their mouth. For the MEP measurement, participants were told to inhale until their lungs were completely filled with air (beginning with the total lung capacity [TLC] point). They then exhaled strongly while holding the device in their lips for 1-2 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jayes L, Haslam PL, Gratziou CG, Powell P, Britton J, Vardavas C, Jimenez-Ruiz C, Leonardi-Bee J; Tobacco Control Committee of the European Respiratory Society. SmokeHaz: Systematic Reviews and Meta-analyses of the Effects of Smoking on Respiratory Health. Chest. 2016 Jul;150(1):164-79. doi: 10.1016/j.chest.2016.03.060. Epub 2016 Apr 19. PMID 27102185
- [Background] Dugral E, Balkanci D. Effects of smoking and physical exercise on respiratory function test results in students of university: A cross-sectional study. Medicine (Baltimore). 2019 Aug;98(32):e16596. doi: 10.1097/MD.0000000000016596. PMID 31393359
- [Background] Gibbs K, Collaco JM, McGrath-Morrow SA. Impact of Tobacco Smoke and Nicotine Exposure on Lung Development. Chest. 2016 Feb;149(2):552-561. doi: 10.1378/chest.15-1858. Epub 2016 Jan 12. PMID 26502117
- [Background] Simmons MS, Connett JE, Nides MA, Lindgren PG, Kleerup EC, Murray RP, Bjornson WM, Tashkin DP. Smoking reduction and the rate of decline in FEV(1): results from the Lung Health Study. Eur Respir J. 2005 Jun;25(6):1011-7. doi: 10.1183/09031936.05.00086804. PMID 15929955
- [Background] Liu JF, Kuo NY, Fang TP, Chen JO, Lu HI, Lin HL. A six-week inspiratory muscle training and aerobic exercise improves respiratory muscle strength and exercise capacity in lung cancer patients after video-assisted thoracoscopic surgery: A randomized controlled trial. Clin Rehabil. 2021 Jun;35(6):840-850. doi: 10.1177/0269215520980138. Epub 2020 Dec 14. PMID 33307766
- [Background] Seo K, Park SH, Park K. Effects of diaphragm respiration exercise on pulmonary function of male smokers in their twenties. J Phys Ther Sci. 2015 Jul;27(7):2313-5. doi: 10.1589/jpts.27.2313. Epub 2015 Jul 22. PMID 26311972